CLINICAL TRIAL: NCT06063720
Title: Prospective Evaluation of Artificial Intelligence-assisted Monitoring of Effective Withdrawal Time on Adenoma Detection
Brief Title: Effective Withdrawal Time and Adenoma Detection Rate
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lui Ka-Luen, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: AIeffectiveV3
Record Dates: First submitted 2023-09-20; First posted 2023-10-02 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Colonic Polyp; Colon Adenoma; Artificial Intelligence
Keywords: Colonic Polyp; Artificial intelligence; Withdrawal time
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AI group: AI monitoring of effective withdrawal time
  Interventions: Device: Endoscreen QC

INTERVENTIONS:
Device: Endoscreen QC — Artificial intelligence monitoring of effective withdrawal time

SUMMARY:
This study prospectively evaluated the role of EWT versus SWT on adenoma detection rate (ADR) and other key quality metrics. In this prospective single-center study, patients undergoing colonoscopy were enrolled. EWT was calculated in real-time using an AI system with endoscopists blinded to the results. We performed multivariable analyses to assess the association of EWT and SWT with binary (e.g., ADR) and count outcomes (e.g., adenoma per colonoscopy [APC]), after adjusting for patient and procedural characteristics.

DETAILED DESCRIPTION:
This was a prospective, single-center observational study designed to determine if an AI-powered metric, Effective Withdrawal Time (EWT), is a superior predictor of colonoscopy quality compared to the traditional Standard Withdrawal Time (SWT). All colonoscopies were performed by qualified endoscopists using high-definition white light video scopes. During the procedure, the scope is first advanced to the start of the large intestine (the cecum). The critical examination phase-the withdrawal-begins as the endoscopist slowly pulls the scope back out, meticulously inspecting the colon lining for abnormalities like polyps. It is during this withdrawal that the key metrics were measured. While SWT is a simple duration timed manually, the AI-measured EWT specifically quantifies the time of high-quality mucosal inspection, automatically excluding periods when the camera view is blurry, obscured, or moving too quickly. A crucial aspect of the methodology was that the endoscopists were blinded to the live EWT measurements to prevent the Hawthorne effect, where individuals alter their behaviour because they are being monitored. The study enrolled adults aged 40 and over, excluding patients with conditions that could confound the findings. The primary goal was to assess the independent impact of EWT on the Adenoma Detection Rate (ADR), a key benchmark based on the detection and removal of precancerous polyps for analysis. To achieve this, researchers used multivariable regression models to isolate EWT's effect from other variables and employed correlation tests to statistically compare whether EWT had a stronger relationship with detection quality than SWT

ELIGIBILITY:
Inclusion Criteria: All adult patients, aged 40 or above, undergoing outpatient colonoscopy will be recruited

Exclusion Criteria:

* history of inflammatory bowel disease
* history of colorectal cancer
* previous bowel resection (apart from appendectomy)
* Peutz-Jeghers syndrome, familial adenomatous polyposis or other polyposis syndromes
* bleeding tendency or severe comorbid illnesses for which polypectomy is considered unsafe.
* Cecum could not be intubated for various reasons
* Poor bowel preparation with Boston Bowel Preparation Scale (BBPS) < 6

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patient will be recruited in Queen Mary Hospital, Hong Kong, China
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rates | During the colonoscopy
  Adenoma detection rates

SECONDARY OUTCOMES:
Polyp detection rate | During that colonoscopy
  Polyp detection rates of the colonoscopy
Serrated lesion detection rate | During colonoscopy
  Serrated lesion detection rates of that colonoscopy
Advanced adenoma detection rate | During colonoscopy
  Advanced adenoma detection rates of that colonoscopy
Adenoma per colonoscopy | During colonoscopy
  Adenoma per colonoscopy
Polyp per colonoscopy | During colonoscopy
  Polyp per colonoscopy
Serrated lesion per colonoscopy | During colonoscopy
  Serrated lesion per colonoscopy
Advanced adenoma per colonoscopy | During colonoscopy
  Advanced adenoma per colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Ka Luen Thomas Lui, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, the University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided